CLINICAL TRIAL: NCT04485897
Title: Can Self-monitoring of the Intraocular Pressure With the Icare HOME Make Hospital-based Diurnal Monitoring Redundant?
Brief Title: Self-monitoring of the Intraocular Pressure Versus Hospital-based Diurnal Monitoring
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 895689
Record Dates: First submitted 2020-07-03; First posted 2020-07-24 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Intraocular Pressure
Keywords: Glaucoma; self-monitoring; intraocular pressure; icare HOME; rebound tonometry
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- icare HOME (Experimental)
  Interventions: Device: icare HOME device (Icare Oy, Vanda, Finland)

INTERVENTIONS:
Device: icare HOME device (Icare Oy, Vanda, Finland) — icare HOME device versus hospital based measurements

SUMMARY:
Glaucoma remains the leading cause of irreversible blindness worldwide. Glaucoma represents a group of diseases that lead to optic nerve damage and corresponding deterioration of the visual field.

Elevated intraocular pressure remains the most important risk factor. Interestingly, glaucomatous damage sometimes occurs despite seemingly normal intraocular pressure.

Recent studies suggest pressure peaks, which are missed under the current practice of spot intraocular measurements during office hours. In order to detect pressure peaks diurnal measurements are mandatory. Costly in-hospital diurnal measurements are the current standard.

The primary study objective is to verify that self-tonometry at home can provide valuable information when looking for pressure peaks in patients with glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Subjects aged 18 and older
* Glaucoma patients and healthy controls
* Best corrected visual acuity >0.1
* Astigmatism ≤ 3dpt.
* Good compliance
* Central corneal thickness (400-650μm)
* Passed certification procedure (detailed description under: Measurements and procedures)
* Therapeutic regimen unchanged throughout the past 30 days

Exclusion Criteria:

* History of ocular trauma
* Corneal condition interfering with tonometry (keratoconus, corneal scaring) Visual acuity <0.1
* Physical or mental disability interfering with self-tonometry (e.g. arthritis, Parkinson's disease)
* Dry eye disease
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-11-26 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of an in- hospital diurnal pressure pattern of intraocular pressure to the pattern derived from self-tonometry using icare HOME in an outpatient setting. | 4 years
  Statistical methods for analysis of continuous method comparison data will be applied. The primary goal is to quantify the extent of agreement between two methods (Intraocular pressure measurement in-hospital and at home) and determine whether they sufficiently agree to be used interchangeably.

SECONDARY OUTCOMES:
variance of diurnal intraocular pressure | 4 years
  Quantitative evaluation of day to day variance of diurnal intraocular pressure measurement in an out-hospital setting in patients with open angle glaucoma, normal tension glaucoma and healthy controls
Influence of daily activities | 4 years
  Influence of daily activities (sports, alcohol and water intake) on intraocular measurements at home (questionnaire)
Change of treatment | 4 years
  Change of treatment due to intraocular pressure peaks during hospitalisation and/or measurements at home

CONTACTS AND LOCATIONS:
Locations (1):
- Cantonal Hospital of Lucerne, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No